CLINICAL TRIAL: NCT06841198
Title: Assessing Cardiovascular Effects: Is There a Time Too Early for Spinal Stimulation in Acute SCI? A Year-Long Evaluation of Autonomic Function Following Injury
Brief Title: Cardiovascular Function and Response to Stimulation Within the First Year After Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Einat Haber, Associate Research Scientist, Kessler Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R1287-25
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries (SCI); Orthostatic Hypotension, Dysautonomic; Cardiovascular; Transcutaneous Spinal Stimulation
Keywords: Transcutaneous Spinal Cord Stimulation; spinal cord stimulation; orthostatic hypotension; blood pressure; cardiovascular; neuromodulation; acute spinal cord injury; chronic spinal cord injury; inpatient rehabilitation; tilt testing; cold pressor test; ambulatory blood pressure monitoring; autonomic dysfunction following spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Shy-Drager Syndrome; Hypotension, Orthostatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: spinal cord transcutaneous stimulation — Stimulation, using the Neostim-5 (Cosyma Ltd.), a 5-channel electrical stimulator, will be administered throughout the study period, beginning shortly after the injury and continuing at regular intervals until one year post-spinal cord injury. It will be performed in two settings:
  1. During seated mapping to identify stimulation sites (potentially T7/8, T11/12, L1/2, and S1/2) and determine stimulation parameters (e.g., frequency, pulse wave, amplitude) that elevate systolic blood pressure (SBP) and maintain it within the target range of 110-120 mmHg.
  2. During 70-degree tilt tests to elicit an orthostatic response (a drop in blood pressure accompanied by symptoms).

SUMMARY:
The study aims to explore how cardiovascular function changes in the first year after a spinal cord injury, and to see how different treatments, like spinal stimulation through the skin (transcutaneous spinal stimulation), affect blood pressure.

The main questions are:

How does stimulation affect blood pressure over the year? What is the level of cardiovascular activation throughout the year?

The study will start during the inpatient stay at the Kessler Institute for Rehabilitation and continue after discharge as an outpatient, totaling about 20-29 sessions over the year.

DETAILED DESCRIPTION:
This clinical study investigates the cardiovascular effects of spinal cord transcutaneous stimulation (scTS) in individuals with recent spinal cord injury (SCI), examining how blood pressure response to stimulation evolves over the first year post-injury. The primary objectives are to determine the optimal timing for initiating scTS for cardiovascular control, characterize blood pressure response evolution to stimulation over one year, and assess autonomic activation patterns through multiple testing methods.

The study will recruit five individuals with recent SCI, specifically targeting those who are 50 days or less post-injury, with an injury level at or above T6, and classified as American Spinal Injury Association Impairment Scale (AIS) A/B. All participants must present with low blood pressure and orthostatic hypotension and be between 18-75 years of age.

The study protocol is divided into inpatient and outpatient phases. During the inpatient phase, consisting of 5-11 sessions, participants undergo a basic assessment including autonomic dysfunction questionnaires, 24-hour blood pressure monitoring, cold pressor testing, and tilt tests with and without stimulation. The protocol also includes 2-3 days of stimulation mapping.

The outpatient phase spans 15-18 sessions over the remainder of the year. Participants undergo monthly mapping sessions and autonomic dysfunction assessments, with comprehensive autonomic testing conducted at 6, 9, and 12 months post-injury. Throughout both phases, researchers perform stimulation mapping across various spinal segments (thoracic, lumbosacral) using a 5-channel electrical stimulator, while monitoring blood pressure and electromyography to target a blood pressure range of 110-120 mmHg.

The study employs multiple assessment tools, including 70° tilt tests with orthostatic symptom evaluation every 5 minutes, cold pressor tests, autonomic dysfunction questionnaires, and 24-hour ambulatory blood pressure monitoring.

The study aims to track primary outcomes including blood pressure response to stimulation at different time points, evolution of orthostatic hypotension symptoms and management, and the pattern of autonomic dysfunction development post-injury.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a spinal cord injury undergoing inpatient rehabilitation at the Kessler Institute for Rehabilitation
* Between 18-75 years old
* 7-50 days after injury
* Injury level ≥ T6 (a cervical or a high-level chest injury)
* Individuals experiencing low blood pressure after the injury
* American Spinal Injury Association Impairment Scale (AIS) A or B

Exclusion Criteria:

* A ventilator is needed for breathing.
* Devices such as brain/spine/nerve stimulators, a cardiac pacemaker/defibrillator, or intra-cardiac lines are present in the body.
* There is a significant disease affecting the blood vessels or signals in the heart, or a recent heart attack (myocardial infarction) has occurred.
* A new medication has been prescribed to treat blood pressure or a heart problem within the last five days (excluding midodrine).
* There is a known infection in the body (e.g., urinary tract infection) or a current illness (e.g., recent diagnosis of deep vein thrombosis (DVT) or other blood clotting issues, and/or a pressure injury that might interfere with the study).
* There is a history of seizures.
* Pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure in seated mapping sessions | The procedure will be repeated throughout the year, starting shortly after the injury and occurring approximately once a month.
  Spatiotemporal mapping sessions involving stimulation of various spinal segments, utilizing different parameters (e.g., frequency, waveform). A BP response in a mapping session will be defined by a significant increase in SBP of at least 20 mmHg with stimulation compared to baseline SBP (without stimulation)
systolic blood pressure in a 70 degree tilt | The procedure will be repeated throughout the year, starting shortly after the injury and occurring approximately every three months
  In this study, tilt-tests are conducted in pairs: first, a standard tilt test (without stimulation), followed by a tilt test with stimulation aimed at preventing orthostatic hypotension. We will compare the drop in systolic blood pressure during the tilt test with stimulation to the drop observed in the standard tilt test.

SECONDARY OUTCOMES:
cold pressor test | The procedure will be repeated throughout the year, starting shortly after the injury and occurring approximately every three months
  In a traditional cold pressor test, the foot is immersed in 0°C ice water, indirectly assessing the degree of sympathetic activation through BP and HR
24-hour ambulatory blood pressure monitoring | The procedure will be repeated throughout the year, starting shortly after the injury and occurring approximately once a month.
  Parameters are recorded automatically every 15 min during the day and every 60 min at night. Participants will be asked to take notes regarding BP-related symptoms, activities, and their time points.
An autonomic dysfunction following spinal cord injury questionnaire | The procedure will be repeated throughout the year, starting shortly after the injury and occurring approximately once a month.
  Assessing the severity and frequency of daily AD and OH episodes and their effect on daily activities

CONTACTS AND LOCATIONS:
Overall Officials: Einat Engel-Haber, MD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
All human subject SCI data will be de-identified. Data shared via a public repository will include demographics (sex, age), injury characteristics (etiology, level and severity of injury), BP measures (systolic, diastolic and heart rate) from mapping, tilt, and 24-hr monitoring data, tilt data (angle, duration, orthostatic questionnaire scores), stimulation data (segment, frequency, amplitude, etc.), responses from the ADF-SCI questionnaire.
Supporting Information: Study Protocol
Time Frame: Upon completing the data collection, the data will be deposited into a public repository for SCI data

REFERENCES:
- [Background] Engel-Haber E, Bheemreddy A, Bayram MB, Ravi M, Zhang F, Su H, Kirshblum S, Forrest GF. Neuromodulation in Spinal Cord Injury Using Transcutaneous Spinal Stimulation-Mapping for a Blood Pressure Response: A Case Series. Neurotrauma Rep. 2024 Sep 20;5(1):845-856. doi: 10.1089/neur.2024.0066. eCollection 2024. PMID 39391052